CLINICAL TRIAL: NCT03248791
Title: Comparison of Two Vasopressor Infusion for Prevention of Post-spinal Hypotension During Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Vasopressor Infusion in Cesarean Delivery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N-86-2017
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Cesarean Section Complications; Spinal Anesthesia
MeSH Terms: interventions — Phenylephrine; Norepinephrine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenylephrine (Active Comparator): Will receive spinal anesthesia using Bupivacaine. Then, phenylephrine infusion by a starting rate of 0.75 mcg/Kg/min. The rate will be then adjusted according to the patient blood pressure
  Interventions: Drug: Phenylephrine; Drug: Bupivacaine
- Norepinephrine (Experimental): Will receive spinal anesthesia using Bupivacaine. Then, norepinephrine infusion by a starting rate of 0.1 mcg/Kg/min. The rate will be then adjusted according to the patient blood pressure
  Interventions: Drug: Norepinephrine; Drug: Bupivacaine

INTERVENTIONS:
Drug: Phenylephrine — Phenylephrine variable infusion with a starting rate of 0.75 mcg/Kg/min.
  Arms: Phenylephrine
Drug: Norepinephrine — Norepinephrine variable infusion with a starting rate of 0.1 mcg/Kg/min.
  Other Names: noradrenaline
  Arms: Norepinephrine
Drug: Bupivacaine — Bupivacaine will be injected in the subarachnoid space with a dose of 10 mg
  Other Names: Marcaine

SUMMARY:
Comparison will be conducted between continuous variable infusions of both drugs (Phenylephrine and Norepinephrine) with starting doses of 0.75 mcg/Kg/min and 0.1 mcg/Kg/min respectively for prophylaxis against Post-spinal hypotension during cesarean delivery.

DETAILED DESCRIPTION:
Maternal hypotension is a common complication after spinal anesthesia for cesarean delivery (CD). Many vasopressors have been used for prevention of post-spinal hypotension (PSH) during CD; however, the optimum protocol for prophylaxis is not established yet. Phenylephrine (PE) is a popular vasopressor used in obstetric anesthesia; however, its use is limited by its marked cardiac depressant nature. Norepinephrine (NE) is a potent vasopressor characterized by both α adrenergic agonistic activity in addition to a weak β adrenergic agonistic activity; thus, NE is considered a vasopressor with minimal cardiac depressant effect; these pharmacological properties would make NE an attractive alternative to PE. In this study, we will compare continuous variable infusion of both drugs (PE and NE) with doses of 0.75 mcg/Kg/min and 0.1 mcg/Kg/min respectively for prophylaxis against PSH during CD.

ELIGIBILITY:
Inclusion Criteria:

* full term
* pregnant women
* scheduled for cesarean section

Exclusion Criteria:

* pre-ecpamsia
* eclampsia
* bleeding
* cardiac dysfuction

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-10 (Estimated)

PRIMARY OUTCOMES:
incidence of post-spinal anesthesia hypotension | 30 minutes after spinal anesthesia
  Defined as the percentage of patients with decreased systolic blood pressure less than 80% of the baseline reading

SECONDARY OUTCOMES:
incidence of severe post-spinal anesthesia hypotension | 30 minutes after spinal anesthesia
  Defined as the percentage of patients with decreased systolic blood pressure less than 60% of the baseline reading
incidence of severe delivery hypotension | 10 minutes after delivery
  Defined as the percentage of patients with decreased systolic blood pressure less than 80% of the baseline reading
systolic blood pressure | 2 hours after subarachnoid block
  systolic blood pressure measured in mmHg
diastolic blood pressure | 2 hours after subarachnoid block
  diastolic blood pressure measured in mmHg
heart rate | 2 hours after subarachnoid block
  number of heart beats per minute
APGAR score | 10 minutes after delivery
  APGAR score of the fetus
incidence of reactive hypertension | 2 hours after spinal anesthesia
  Defined as the percentage of patients with increased systolic blood pressure more than 80% of the baseline reading

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Professor, Study Director — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No